CLINICAL TRIAL: NCT04526418
Title: Evaluation of the 24/7 EEG SubQ System for Ultra Long-Term Recording of Patients With Epilepsy Involving the Temporal Lobe Region. An Open-label, Prospective, Paired, Comparative Study.
Brief Title: Evaluation of the 24/7 EEG SubQ System for Ultra Long-Term Recording of Patients With Epilepsy Involving the Temporal Lobe Region.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility analysis reached
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U002
Record Dates: First submitted 2020-08-10; First posted 2020-08-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
Keywords: Ultra Long-Term Recording of Patients with Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: open-label, prospective study with a paired comparative design for pivotal evaluation of the safety and effectiveness of the 24/7 EEC SubQ system in subjects with epilepsy involving the temporal lobe region.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- 24/7 EEG™ SubQ System (Experimental): To demonstrate the electrographic seizure recording effectiveness of the 24/7 EEG™ SubQ system by comparison to simultaneous inpatient video-EEG data.
  Interventions: Device: 24/7 EEG™ SubQ system

INTERVENTIONS:
Device: 24/7 EEG™ SubQ system — Electrographic seizure recording sensitivity of an ipsilaterally implanted 24/7 EEG™ SubQ system: proportion of identified ipsilateral seizures as compared to ipsilateral video-EEG during admission to the Epilepsy Monitoring Unit

SUMMARY:
The 24/7 EEG™ SubQ system will be compared to simultaneously recorded video-EEG in the Epilepsy Monitoring Unit (gold standard) and to self-reported seizure log books throughout 12 weeks of outpatient EEG recording.

The present study is a 12-week open-label, prospective study with a paired, comparative design for pivotal evaluation of the safety and effectiveness of the 24/7 EEGTM SubQ system in subjects with epilepsy involving the temporal lobe region .

2-5 sites in Europe Up to 10 sites in US

ELIGIBILITY:
INCLUSION CRITERIA

1. Subject is 18-75 years old.
2. Semiology of seizures compatible with temporal lobe involvement.
3. Paraclinical findings supporting temporal seizure involvement. Such proof may consist of: - previous EEG recording interpreted as compatible with temporal involvement OR - radiological findings demonstrating pathology in the temporal area (CT, MRI, FDG-PET or SPECT).
4. Uncontrolled epileptic seizures.
5. Subject has planned clinical EMU admission with an admission goal including capturing epileptic seizures, within 12 weeks after the date of UNEEG™ SubQ implant.
6. Subject is willing and able to provide written informed consent.
7. Subject is able to complete all study-required procedures, assessments and follow-up.

EXCLUSION CRITERIA

1. Subject has a condition that places him/her at a high at high risk of surgical complications, such as an active systemic infection or a hemorrhagic disease.
2. Subject receives frequent (more than 2 days per week) treatment with drugs of the following types:

   1. antiplatelets
   2. anticoagulants
   3. chemotherapeutics
   4. non-steroid anti-inflammatory drugs (NSAID)
3. Subject has skeletal deformities or damage at the proposed implantation site to an extent that impedes correct electrode placement.
4. Subject is involved in therapies with other active implantable devices that deliver electrical energy above the clavicular area, such as implantable brain stimulation, external/transcranial brain stimulation, vagus nerve stimulator (VNS) and cochlear implant(s).
5. Subject is pregnant
6. Subject has contraindicated profession or hobby
7. Subject is scheduled to undergo contraindicated treatments/investigations
8. Infection at the implant site
9. Subject has contraindication to the use of anesthetic used for in/ex plantation.
10. Subject is unable to use/operate the device system
11. Subject has abnormal Laboratory findings as follows:

    * Serum creatinine ≥ 3 times upper reference value
    * Alanine aminotransferase (ALT), alkaline phosphatase or bilirubin ≥ 3 times upper reference value
    * Activated Partial Thromboplastin Time (APTT) > 50 seconds
    * thrombocyte count < 50 or >1000 x 109/L
    * International Normalised Ratio (INR) ≥ 1.6
    * Any other clinical or paraclinical finding that in the opinion of the Investigator would interfere with participation in the study or would confound interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
number of seizures | comparasion in EMU for 3-14 days period, where patients are hospitalized.
  numbers of seizures as detected in EEG data from SubQ to be compared with number of seizures detected in golden standard (video EEG).

SECONDARY OUTCOMES:
adverse event | 2 years
  safety reporting

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gelfand, Principal Investigator — University of Pennsylvania
Locations (12):
- United States (9):
  - University of California, Los Angeles, California
  - University of South Florida (USF) Neurology Department, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack Meridian Health, Neptune City, New Jersey
  - Northwell Health Department of Neurosurgery, Great Neck, New York
  - Cleveland Clinic, Neurological Institute, Cleveland, Ohio
  - University of Pennsylvenia, Philadelphia, Pennsylvania
  - UT Health Houston, Houston, Texas
- Hopital Erasme - Universite Libre de Bruxelles, Brussels, Belgium
- Germany (2):
  - Krankenhaus Mara, Gesellschaft für Epilepsieforschung e.V., Bielefeld
  - Universität Klinikum Freibrug, Freiburg im Breisgau

IPD SHARING:
Plan to Share IPD: No